CLINICAL TRIAL: NCT03933683
Title: Indirect Non-invasive Evaluation of Pudendal Neuropathy by Dynamic Transperineal Ultrasound in Patients With Pelvic Floor Dysfunction
Brief Title: Indirect Non-invasive Evaluation of Pudendal Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Luigi Brusciano, Clinical Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 229/19
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; pudendal neuropthy; pudendal nerve terminal motor latency
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pathologic Group: Patients affected by Fecal Incontinence
  Interventions: Device: Pudendal nerve terminal motor latency assessment
- Control Group: Healty volunteers cohort
  Interventions: Device: Pudendal nerve terminal motor latency assessment

INTERVENTIONS:
Device: Pudendal nerve terminal motor latency assessment — After a specialized coloproctology evaluation, each patient with pelviperineal dysfunction was addressed to dynamic transperineal ultrasound to determine anterior and posterior displacement of puborectalis muscle, and subsequently a blinded neurophysiologist performed pudendal nerve terminal motor latency assessment to identify pudendal neuropathy.
  Other Names: Dynamic transperineal Ultrasound

SUMMARY:
Purpose: Pelvic floor is a complex anatomical entity and its neuromuscular assessment is evaluated through electromyography, evoked potentials and pudendal nerve terminal motor latency. An innovative approach is the study of pelvic floor through dynamic transperineal ultrasound (DTU). The aim of this study is to evaluate if anterior and posterior displacement of puborectalis muscle, studied by DTU, is a feasible and effective method to diagnose pudendal neuropathy alternatively to conventional St. Marks' glove.

Methods:Patients affected by fecal incontinence (FI) addressed to our referral center of coloproctology at University of Campania were prospectively assessed. After a specialized coloproctology evaluation, each patient with pelviperineal dysfunction was addressed to DTU to determine anterior and posterior displacement of puborectalis muscle, and subsequently a blinded neurophysiologist performed pudendal nerve terminal motor latency assessment to identify pudendal neuropathy. In order to compare the data, a cohort of 34 healthy volunteers was enrolled.

DETAILED DESCRIPTION:
This study is reported according to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement for cohort studies. Between January 2008 and December 2016, female patients affected by fecal incontinence (FI) or urinary incontinence referred to our referral center of coloproctology (master of pelvi-perineal rehabilitation and master of coloproctology) at University of Study of Campania "Luigi Vanvitelli" of Naples were prospectively assessed. Inclusion criteria were age ≥16 and symptoms of faecal incontinence or constipation. Exclusion criteria were past history of anorectal or vaginal surgery, history of pelvic radiation or tumors and inability to complete the study protocol. Patients with pelviperineal dysfunction were enrolled in the study (Group A). Clinical symptoms were graded as follows: constipation was evaluated according to the Wexner Scale (0-30), continence was evaluated according to Cleveland Clinic incontinence score (0-20)13-14. The following information were collected: age, symptoms, grading, previous pelvic surgery. In order to compare and analyse the data, a cohort of 34 healthy volunteers was enrolled among students and residents of University of Campania "Luigi Vanvitelli" (Group B). The local ethical committee approved the study protocol.

Patients All patients were assessed during a specialized coloproctology evaluation in our teaching Hospital. A clinical examination was performed in all patients and information on bowel function, pregnancies, episiotomy, previous surgery and associated diseases were recorded. A preoperative informed consent was acquired in every case and the physicians explained to the patients the details and the aims of the procedures.

Each patient underwent a DTU by an expert coloproctologist (LB) with great experience of perineal ultrasonography, person in charge of a master of coloproctology and of master of pelvi-perineal rehabilitation at University of Study of Campania "Luigi Vanvitelli" of Naples. Subsequently, all patients underwent PNTML evaluation using the St. Marks glove mounted pudendal nerve stimulator (St. Mark's 13 L40® Dantec Elektronic, Skovlunde, Denmark), performed by a blinded neurophysiologist (FT).

Dynamic Transperineal Ultrasound Voluntary contraction of the perineum and of the PR muscle leads to a shortening of the PR muscle itself. The anal canal moves in the direction of the pubic bone and diminishes the anorectal angle. In contrast, relaxation of the PR muscle, which occurs while attempting defecation, lengthens the PRS and opens the anorectal angle. Contraction and relaxation of the PR muscle can be measured with DTU. DTU, in fact, is a morphological and functional procedure assessing puborectal function. It is cheap, feasible, well tolerated and reproducible. The patient is placed in the dorsal lithotomy position, with hips flexed and abducted, and a 3-6 MHz conventional convex transducer and field of view at least 70° positioned on the perineum between the mons pubis and the anal margin. In the mid-sagittal plane, all anatomical structures (bladder, urethra, vaginal walls, anal canal and rectum) between the posterior surface of the symphysis pubis and the posterior part of the levator ani are visualized3. [Figure 1] The probe is progressively inclined until the anal sphincter is visible. Changing application pressure and probe inclination, allows to scan the entire anal canal in transversal section. After the sphincter identification, a further longitudinal image obtained with a 90° rotation of the scanning plane allows to observe the PR sling behind the rectum.

The first caliper is placed on the anterior border of the PR in resting position; the second one is placed on the anterior border of PR in straining or squeezing position in order to respectively obtain the measure AD or the PD.

In healthy patients, the AD should be more than 7mm during squeezing and the PD more than 6mm, during straining.

Pudendal nerve terminal motor latency Pudendal nerve terminal motor latency is an affordable technique to evaluate anal sphincter innervation; it reflects the conduction velocity of the fastest motor nerve fiber supplying the anal sphincter.

In order to execute the examination a glove-mounted electrode (St. Mark's 13 L40® Dantec Elektronic, Skovlunde, Denmark) is used to measure pudendal nerve conduction time.

It is inserted into the anal canal with patients laying in Sims position. Both right and left pudendal nerves are stimulated using a pulse of 50 V, for 0.1 ms at a rate of 1 pulse per second over the ischial spines until a reproducible latency is obtained.

We selected the shortest reproducible latency recorded for each patient according to the neurophysiologist opinion. Prolonged PNTML was defined as greater than or equal to 2.2 ms.

ELIGIBILITY:
Inclusion Criteria:

* age ≥16
* symptoms of faecal incontinence

Exclusion Criteria:

* past history of anorectal or vaginal surgery
* history of pelvic radiation or tumors -inability to complete the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients affected by fecal incontinence (FI) or urinary incontinence to our referral center of coloproctology (master of pelvi-perineal rehabilitation and master of coloproctology) at University of Study of Campania "Luigi Vanvitelli" of Naples were prospectively assessed.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Concordance between pudendal nerve motor latency and dynamic transperineal ultrasound for the evaluation of pudendal neuropathy | 3 months
  Concordanace between pudendal nerve terminal motor latency (the actual gold standard in the evaluation of pudendal neuropathy, expressed in ms) and puborectalis displacement (expressed in mm) analysed by dynamic transperineal ultrasound for the evaluation of pudendal neuropathy in gruop of patients affected by fecal incontince. The data will be compared to the results obtained in a cohort of healty volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Brusciano, Prof, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Derived] Brusciano L, Gambardella C, Roche B, Tolone S, Romano RM, Tuccillo F, Del Genio G, Terracciano G, Gualtieri G, Docimo L. Dynamic transperineal ultrasonography correlates with prolonged pudendal nerve latency in female with fecal incontinence. Updates Surg. 2020 Dec;72(4):1187-1194. doi: 10.1007/s13304-020-00838-y. Epub 2020 Jun 28. PMID 32596803